CLINICAL TRIAL: NCT01788839
Title: Longitudinal Sexual and Reproductive Health Study of Women With Breast Cancer and Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 12-249
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Lymphoma; Hodgkin's Lymphoma
Keywords: Sexual and Reproductive Health; premenopausal; postmenopausal; 12-249; Fertility
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Hodgkin Disease; Coitus | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood draw

GROUPS / COHORTS (2):
- women with breast cancer: This study is a prospective, observational, longitudinal study assessing the prevalence of sexual dysfunction and distress in premenopausal and postmenopausal women with breast cancer. This study will also evaluate the severity, time course, and predictors of sexual dysfunction. Breast cancer patients and survivors will be administered surveys of comprehensive questionnaires related to sexual function. In the case that participants miss the follow up questionnaires, study staff may contact the patient by phone to request and record the patients" responses. The study staff may also mail the missed questionnaires to each patient.
  Interventions: Behavioral: surveys; Other: Blood draw; Device: Transvaginal ultrasounds
- women with lymphoma: This study is a prospective, observational, longitudinal study assessing the prevalence of sexual dysfunction and distress in premenopausal and postmenopausal women with Diffuse Large B-cell Lymphoma or Hodgkin's Lymphoma. This study will also evaluate the severity, time course, and predictors of sexual dysfunction. Lymphoma patients and survivors will be administered surveys of comprehensive questionnaires related to sexual function. In the case that participants miss the follow up questionnaires, study staff may contact the patient by phone to request and record the patients" responses. The study staff may also mail the missed questionnaires to each patient.
  Interventions: Behavioral: surveys; Other: Blood draw; Device: Transvaginal ultrasounds

INTERVENTIONS:
Behavioral: surveys — A survey including the Female Sexual Function Index (FSFI), the Modified Female Sexual Function Index (FSFI-M), the Modified Female Sexual Function Index Follow-Up (FSFI-M Follow-Up) the Sexual Activity Questionnaire (SAQ), the Female Sexual Distress Scale (FSDS-R), the Menopausal Symptom Check List (MSCL), Patient-reported Outcomes Measurement Information System Sexual Function Instrument (PROMIS-SF), Abbreviated Dyadic Adjustment Scale for Relationships (ADAS), Reproductive Health Survey-baseline (RHS-B). Reproductive Health Survey-followup and (RHS-F1)Reproductive Health Survey-followup (RHS-F2) will be conducted at the following intervals: baseline/before chemotherapy +/- 1 month, 3 months after baseline +/- 1 month, 6 months after baseline +/- 1 month, 1 year after baseline +/- 1 month, and at intervals during survivorship that include yearly for 5 years +/- 2 months.
Other: Blood draw — Those patients receiving chemotherapy who consent to the optional blood draw will provide blood at baseline (before start of chemotherapy), 12 months after baseline (+/-1 month) and 24 months after baseline (+/-2 months). All patients in the subset of the premenopausal cohort receiving tamoxifen only will have required blood draws at baseline (before they begin taking tamoxifen), at 6 months post-baseline/start of tamoxifen (+/- 2 weeks), 12 months post-start of tamoxifen (+/-1 month) and 24 months post-start of tamoxifen (+/-2 months). We will ask these participants for blood draws on day 1, 2, 3 or 4 of their menses at baseline and 6 months post-baseline/start of tamoxifen and during months 1 through 5 post-baseline/start of tamoxifen.
Device: Transvaginal ultrasounds — Transvaginal ultrasounds are used to determine the number of antral follicles in each ovary. They will be performed to evaluate both the number and size of antral follicles of premenopausal women on Tamoxifen as antral follicle count is a good predictor of ovarian reserve and response. All patients in the subset of the premenopausal cohort receiving tamoxifen only will also have required transvaginal ultrasounds at baseline (before they begin taking tamoxifen) and at 6 months post-start of tamoxifen (+/- 2 weeks).

SUMMARY:
The purpose of this study is to see how cancer treatment affects sexual and reproductive function. The patient will also be asked to participate in blood draws to see if and how cancer treatment affects the ovaries and the ability to have children (fertility). These blood draws are optional and the patient can still participate in the questionnaire portion of the study even if they choose not to have their blood drawn.

ELIGIBILITY:
Inclusion Criteria:

Subject Inclusion Criteria for Cohort of Premenopausal Women with Early Stage Breast Cancer and Lymphoma

* Women, 18 years of age and older
* Premenopausal women at time of diagnosis who have either been pregnant or had at least one menstrual period in the last 12 months

  * Note: premenopausal women at time of diagnosis who have not been pregnant or have not had at least one menstrual period in the last 12 months are able to participate only if they have had an intrauterine device (IUD) in place within the last 12 months.
* Women with newly diagnosed breast cancer (stage 0-III) who are within 1 month of starting systemic treatment or women with any aggressive lymphoma being treated with first line therapy with curative intent.
* Breast cancer patients with any receptor type
* English speaking
* Able to participate in the informed consent process

Subject Inclusion Criteria for Tamoxifen Only Subset of Cohort of Premenopausal Women with Early Stage Breast Cancer and Lymphoma

* Women, 18 years of age and older.
* Premenopausal women at time of diagnosis who have either been pregnant or had at least one menstrual period in the last 12 months

  * Note: premenopausal women at time of diagnosis who have not been pregnant or have not had at least one menstrual period in the last 12 months are able to participate only if they have had an intrauterine device (IUD) in place within the last 12 months.
* Women with newly diagnosed breast cancer (stage 0-III) who have not yet started treatment and are planning to start Tamoxifen as their only form of systemic treatment within one month
* Breast cancer patients with any receptor type
* English speaking
* Able to participate in the informed consent process

Subject Inclusion Criteria for Cohort of Postmenopausal Women with Early Stage Breast Cancer and Lymphoma

* Women, 18 years of age and older.
* Postmenopausal women at time of diagnosis who have been without period for ≥ 2 years.
* Women with newly diagnosed breast cancer (stage 0-III) who are within 1 month of starting systemic treatment or women with any aggressive lymphoma being treated with first line therapy with curative intent.
* Breast cancer patients with any receptor type
* English speaking
* Able to participate in the informed consent process

Exclusion Criteria:

Subject Exclusion Criteria for both Pre and Postmenopausal Women with Early Stage Breast Cancer and Lymphoma

* Active secondary cancer requiring cytotoxic chemotherapy
* Prior systemic treatment for a malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women for both the premenopausal and postmenopausal cohorts diagnosed with stage 0-III breast cancer or any aggressive lymphpoma will be recruited from breast cancer and lymphoma clinics.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2013-02; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
determine the natural history of sexual and reproductive health | 5 years

SECONDARY OUTCOMES:
predictors of sexual dysfunction during and after treatment | 5 years
impact of treatment on self-reported future pregnancy/reproductive health | 5 years
factors that influence decisions regarding fertility preservation | 5 years
  Before treatment and family building after treatment
comparison of sexual function between breast cancer and lymphoma patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/